CLINICAL TRIAL: NCT03525327
Title: USC Choreographic Institute Line Dance Study
Brief Title: University of Southern California Choreographic Institute Line Dance Study
Acronym: USCCILDS
Status: Completed | Type: Observational
Sponsor: Patrick Corbin (Other)
Responsible Party: Sponsor-Investigator, Patrick Corbin, Assistant Professor of Practice, University of Southern California
Organization: University of Southern California (Other)
Other Study IDs: UP-17-00676
Record Dates: First submitted 2017-10-31; First posted 2018-05-15 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Quality of Life
Keywords: Dance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Line Dance Class participants: The group will be participating in line dance classes as intervention.
  Interventions: Other: Line Dance Class

INTERVENTIONS:
Other: Line Dance Class — Line or party dances to be taught will include:
  Electric Slide (Mainland USA)Hukilau (Hawaii)Cupid Shuffle (Mainland USA)Poco Poco (Philippines)Cha Cha Slide (Mainland USA)Tush Push (Mainland USA)Trojan Crawl (Mainland USA)Wobble (Mainland USA)Goyang Maumere (Indonesia)

SUMMARY:
This study will include dance protocols for targeted therapeutic interventions measuring the effect of line dancing on cognitive, emotional and social well-being. The hypothesis is that participating in a one-hour line dance class once a week for twelve weeks will decrease stress levels and enhance participants' quality of life, as measured by interview survey questionnaires. Questionnaires will be administered at the beginning, mid-point, and end of the study. The objectives of the study are threefold: to quantify the beneficial effects of line dancing on quality of life including cognitive, emotional and social well-being; to identify how non-lifetime, amateur dance practitioners can benefit from dancing; and to demystify dance class and make it accessible to people who are not interested in learning a specific dance technique or concert/art dance. Line dancing is a cross-cultural, intergenerational activity that could fill this role.

DETAILED DESCRIPTION:
Synchronous movement to music (dance) is an essential aspect of human experience. Groups of people historically engage in dance in social situations where bonding is important. For example, dance is a common activity at parties, weddings, funerals, and other ritualistic or religious ceremonies.

In line or party dances, dancers learn through wireless transmission or simple synchrony. By mimicking the leader's movements in time with the music, the group learns the dance and experiences the same dyadic relationship as children experience learning with a parent. Although it is taking place in a group setting the dyadic relationship is no less intimate or mysterious. The wireless transmission creates a non-verbal bond based on trust. The group trusts that the leader is going to share information that is going to be fun and psychically nourishing. The leader tends to the group with care and confidence, instilling in the group a sense of security and calm.

This study will include dance protocols for targeted therapeutic interventions measuring the effect of line dancing on cognitive, emotional and social well-being. The hypothesis is that participating in a one-hour line dance class once a week for twelve weeks will decrease stress levels and enhance participants' quality of life, as measured by interview survey questionnaires. Questionnaires will be administered at the beginning, mid-point, and end of the study. The objectives of the study are threefold: to quantify the beneficial effects of line dancing on quality of life including cognitive, emotional and social well-being; to identify how non-lifetime, amateur dance practitioners can benefit from dancing; and to demystify dance class and make it accessible to people who are not interested in learning a specific dance technique or concert/art dance. Line dancing is a cross-cultural, intergenerational activity that could fill this role.

This twelve-week line dance course takes place at the Ahmanson Senior Center at the Expo Center adjacent to University of Southern California University Park Campus. Nineteen senior citizen participants have agreed to participate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be between the gaes of 50 and 90 years old.

Exclusion Criteria:

* Younger than 50 or older than 90.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the Ahmanson Senior Center
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF | Change is being assessed from baseline measure at week 1 to last meeting at six-months.
  The World Health Organization Quality of Life Questionnaire short form

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Corbin, MFA, Principal Investigator — Faculty Lead
Locations (1):
- Ahamnson Senior Center at Expo Center, Los Angeles, California, United States